CLINICAL TRIAL: NCT06539793
Title: Effect of Neuromodulation on Pain Biomarkers and Functional Outcome in Patients With Fibromyalgia Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Alshimy (Other)
Responsible Party: Sponsor-Investigator, Ahmed Alshimy, Lecturer and Consultant in Physical Therapy at Department of Neurology and it's Surgery. Faculty of Physical Therapy Al Ryada University for Science and Technology, Egypt, AlRyada University for Science & Technology
Organization: AlRyada University for Science & Technology (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005277
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia; NEUROMODULATION; Centralization; PAIN BIOMARKERS; FUNCTIONAL OUTCOME
MeSH Terms: conditions — Fibromyalgia | interventions — Exercise; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (A) (Experimental): Patients will receive exercises, and sham Non-Invasive Neuromodulation, 3 sessions per week (one hour for each session) for 4 weeks.
  Interventions: Other: Aerobic Exercises; Other: Transcutaneous electrical nerve stimulation
- Control group (B) (Experimental): Patients will receive exercises as in group (A) in addition to Non-Invasive Neuromodulation 3 sessions per week (one hour for each session) for 4 weeks.
  Interventions: Other: Aerobic Exercises

INTERVENTIONS:
Other: Aerobic Exercises — Treadmill 20 minutes including 5 minutes warm up and 5 minutes cool.
Other: Transcutaneous electrical nerve stimulation — will be applied for all patients, which uses an asymmetrical biphasic alternating current in the continuous mode (pulse duration 100 µs, low frequency). TENS intensity will increase slowly, and patients will be instructed to indicate sensory threshold (ST); then, the intensity are going to increase until the sensation perceived as "strong but comfortable" (SC1). The duration will be for 30 minutes, 3times/ week for 4 weeks
  Arms: Study group (A)

SUMMARY:
Fibromyalgia is the third most common musculoskeletal condition in terms of prevalence, after lumbar pain and osteoarthritis. Its prevalence is around 2-4 % and is more frequent in women than in men; the prevalence is highest in age the range of 40-60 years.

DETAILED DESCRIPTION:
Group A (Control Group): Patients will receive exercises, and sham Non-Invasive Neuromodulation, 3 sessions per week (one hour for each session) for 4 weeks.

Group B (Study Group): Patients will receive exercises as in group (A) in addition to Non-Invasive Neuromodulation 3 sessions per week (one hour for each session) for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients fibromyalgia from both genders.
2. The duration of fibromyalgia is more than 6 month (all patients with history of cervical or lumbar pain) and following diagnosis of FM using the 2016 revised FM criteria, on the basis of the ACR-2010 criteria.
3. Their ages will be ranged from 25-35 years old.
4. They will be medically stable and have sufficient cognitive abilities that enable them to understand and follow instruction according to Montreal Cognitive Assessment (MoCA) >26.

Exclusion Criteria:

1. Other Neurological diseases as stroke , multiple sclerosis, Parkinson's disease and motor neuron disease
2. Pacemaker
3. Spinal fusion-cervical or lumbar
4. Metal implants in the spine
5. Pregnancy
6. Epilepsy
7. Severe psychiatric disorder or alcohol and drug abuse.
8. Unstable medical condition which could compromise the participant's welfare or confound the study results.
9. Uncontrolled blood pressure or diabetes
10. Visual or auditory problems.
11. Active inflammatory conditions

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-04-04 (Estimated); Study Completion 2025-07-03 (Estimated)

PRIMARY OUTCOMES:
Pain Numeric Pain Rating Scale | 4 weeks
  Assessment of pain intensity (0-no pain, 10-most intense pain)
Biochemical analysis | 4 weeks
  Assessment of pain intensity through the change of blood cortisol level, plasma cytokine level, antinuclear antibody (ANA) level. Blood samples will be taken between the hours of 08:00-09:00 in the morning. Two blood samples will be taken from the patients before and after treatment.
Fibromyalgia Impact Questionnaire | 4 weeks
  Assess functional outcome
Pressure Pain Thresholds | 4 weeks
  Assess pain sensitivity through pressure algometer

CONTACTS AND LOCATIONS:
Locations (1):
- Al Ryada University for Science and Technology, Sadat, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No